CLINICAL TRIAL: NCT04327011
Title: A Continuation Protocol for Patients Previously Enrolled in a Study of Toca 511
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Tocagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tg 511-09-01
Record Dates: First submitted 2016-12-21; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Glioblastoma Multiforme; Astrocytoma; Gliomas, Malignant
Keywords: glioma; glioblastoma; glioblastoma multiforme; Grade IV astrocytoma; brain cancer; recurrent glioblastoma; GBM; AA; AOD; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic oligoastrocytoma; high grade glioma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Glioma; Brain Neoplasms; Oligodendroglioma | interventions — vocimagene amiretrorepvec; Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Single arm Toca 511 vector/5-FC prodrug
  Interventions: Biological: Toca 511 vector; Drug: Toca FC • Flucytosine • 5-FC • 5-Fluorocytosine

INTERVENTIONS:
Biological: Toca 511 vector — Toca 511 consists of a purified retroviral replicating vector encoding a modified yeast cytosine deaminase (CD) gene. The CD gene converts the antifungal 5-flurocytosine (5FC) to the anticancer drug 5-FU in cells that have been infected by the Toca 511 vector
  Other Names: vocimagene amiretrorepvec; RRV; retroviral replicating virus
Drug: Toca FC • Flucytosine • 5-FC • 5-Fluorocytosine — Toca FC is an extended-release formulation of flucytosine.
  Other Names: Extended Release 5-FC; 5-FC; 5-Fluorocytosine

SUMMARY:
This is a multicenter, open-label, continuation study to allow subjects who have previously received Toca 511 to continue to receive Toca FC and to allow for extended safety observations. Subjects will be seen on an every six week basis for 1 year or longer. Subjects who continue to receive Toca FC will receive the dose described in the "parent" protocol. If the Toca FC dose is adjusted for any reason, the serum concentration will be monitored. Gadolinium (Gd)-enhanced magnetic resonance imaging (MRI) scans will be performed as per standard of care.

If the subject has recurred/progressed, repeat intracranial injection of Toca 511 followed by Toca FC treatment may be offered to consenting patients.

Subjects who enter the study to continue Toca FC and subsequently discontinue Toca FC, and subjects who are only willing or able to perform limited testing will have viral testing alone, at the appropriate intervals.

After the first year, subjects will be seen twice yearly for the next 4 years and then contacted yearly for the next 10 years.

All subjects will be followed on study for at least 5 years regardless of whether they are taking Toca FC.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form
* Subject received Toca 511 in prior study.
* Subject is willing to abide by protocol

Exclusion Criteria:

* Subject has history of allergy or intolerance to flucytosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Long term safety follow up | From study entry up to 15 years
  This will be based on treatment emergent adverse events, clinical laboratory values and viral testing.

SECONDARY OUTCOMES:
Overall survival in days from the initial Toca 511 administration on parent study to the date of death. | From initial Toca 511 administration to death of last patient alive for up to 15 years.

OTHER OUTCOMES:
Progression-free survival in days from the initial Toca 511 administration on parent study to confirmed disease progression or death from any cause. | from initial toca 511 administration to time of progression or death of any cause for up to 15 years.
Objective response rate from initial dose of Toca FC from the parent protocol | Time from initial dose of Toca FC to death of last patient alive for up to 15 years.

CONTACTS AND LOCATIONS:
Overall Officials: Asha Das, MD, Study Director — Tocagen Inc.; Michael Vogelbaum, MD, PhD, NS, Principal Investigator — The Cleveland Clinic
Locations (11):
- United States (11):
  - University of California, Los Angeles, Los Angeles, California
  - UCSD, San Diego, California
  - UCSF, San Francisco, California
  - Henry Ford Health System, Detroit, Michigan
  - JFK Medical Center Neuroscience Institute, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University, Hackensack, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No